CLINICAL TRIAL: NCT01856907
Title: A Randomized Pilot Study Evaluating Combination Dipeptidyl Peptidase-4 Inhibitor Sitagliptin Plus Metformin Compared to Metformin Monotherapy and Placebo on Metabolic Abnormalities in Women With a Recent History of GDM
Brief Title: Sitagliptin + Metformin Compared to Metformin Monotherapy and Placebo in Women With a Recent GDM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Woman's (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Karen Elkind-Hirsch, Director of Research, Woman's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RP13-009
Record Dates: First submitted 2013-05-14; First posted 2013-05-20 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Disorder of Glucose Regulation
Keywords: prediabetes; impaired fasting/impaired glucose tolerance; post gestational diabetes; diabetes prevention
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Metformin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitagliptin-Metformin (Experimental): 50 mg/1000 mg twice a day (BID)
  Interventions: Drug: Sitagliptin-Metformin
- Placebo pill (Placebo Comparator): 1 pill/BID for 16 weeks
  Interventions: Drug: Placebo pill
- Metformin (Active Comparator): 1000 mg BID
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Sitagliptin-Metformin — Experimental -dipeptidyl peptidase-4 (DPP-4) inhibitor- oral medication
  Other Names: Janumet
  Arms: Sitagliptin-Metformin
Drug: Metformin — Biguanide- insulin sensitizer
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo pill — Will evaluate effect of lifestyle and diet only
  Other Names: placebo control
  Arms: Placebo pill

SUMMARY:
Gestational diabetes mellitus (GDM) is defined as "any degree of glucose intolerance with onset or first recognition during pregnancy." GDM is one of the most frequent metabolic disorders occurring during pregnancy. Approximately 7% of all pregnancies in the United States are complicated by gestational diabetes resulting in more than 200,000 cases annually. There is epidemiologic evidence associating GDM with insulin resistance, glucose intolerance, and type 2 diabetes (DM2). Among all the risk factors of diabetes mellitus, the experience of gestational diabetes is the strongest one. Systematic reviews of older studies conclude that 35-60% women with gestational diabetes will develop type 2 diabetes at rates much greater than control groups who did not have glucose intolerance during pregnancy. Studies are needed for optimal postpartum and long-term health of women who have had GDM. Recent evidence suggests that incretin-based therapies may be useful for the treatment of DM2 because continuous administration of glucagon-like peptide 1 (GLP-1) produces substantial improvements in glucose control and ß-cell function in subjects with DM2. Inhibition of dipeptidyl peptidase-4 (DPP-4) increases the concentration of GLP-1 and may potentially delay disease progression in GDM considering the ß-cell function improvement in DM2 and ß-cell mass shown to increase in animal models. This study will examine if combination sitagliptin (a DPP-4 inhibitor)-plus metformin is more effective than metformin alone or placebo in improving metabolic parameters, specifically the impact on β-cell function, in prior GDM women with glucose abnormalities.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is defined as "any degree of glucose intolerance with onset or first recognition during pregnancy." GDM is one of the most frequent metabolic disorders occurring during pregnancy. Approximately 7% of all pregnancies in the United States are complicated by gestational diabetes resulting in more than 200,000 cases annually. There is epidemiologic evidence associating GDM with insulin resistance, glucose intolerance, and type 2 diabetes (DM2). Among all the risk factors of diabetes mellitus, the experience of gestational diabetes is the strongest one.

Gestational diabetes is often the culmination of years of unrecognized and unmodified diabetes risk factors that lead to overt and occult clinical manifestations during pregnancy. Systematic reviews of older studies conclude that 35-60% women with gestational diabetes will develop type 2 diabetes at rates much greater than control groups who did not have glucose intolerance during pregnancy. The higher rates were in studies of particular ethnic groups in the U.S. Presently, in the literature, there are described new, more efficient methods of diabetes prevention in groups with a high risk of this disorder, which involve both, lifestyle modification and pharmacological therapies. Lifestyle intervention was found to reduce the incidence of type 2 diabetes by 58% and metformin by 31% as compared with placebo. Studies are needed for optimal postpartum and long-term health of women who have had GDM. Considerable recent evidence suggests that incretin-based therapies may be useful for the treatment of DM2 because continuous administration of glucagon-like peptide 1 (GLP-1) produces substantial improvements in glucose control and ß-cell function in subjects with type 2 diabetes. Inhibition of dipeptidyl peptidase-4 (DPP-4) increases the concentration of GLP-1 and may potentially delay disease progression in GDM considering the ß-cell function improvement in DM2 and ß-cell mass shown to increase in animal models. This study will examine if combination sitagliptin-plus metformin is more effective than metformin alone or placebo in improving metabolic parameters, specifically the impact on β-cell function, in at-risk women with a recent history of GDM.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years to 42 years of age who experienced gestational diabetes mellitus (GDM) during recent (within 12 months) pregnancy with prediabetic hyperglycemia determined by an oral glucose tolerance test (OGTT) with 75 g glucose postpartum. Study subjects will be inclusive of prior GDM women with impaired fasting glucose (IFG), impaired glucose tolerance (IGT), or both (IFG/IGT) postpartum.
* Written consent for participation in the study

Exclusion Criteria:

* Cholestasis during the past pregnancy
* Any hepatic diseases in the past (viral hepatitis, toxic hepatic damage, jaundice of unknown etiology)
* Serum aspartate transaminase (AST) and/or alanine aminotransferase (ALT) level exceeding more than twice normal lab values
* Presence of hypersensitivity to sitagliptin or other DPP-4 inhibitor
* Current use of metformin, thiazolidinediones, GLP-1 receptor agonists, DPP-4 inhibitors, or weight loss medications (prescription or over the counter [OTC])
* Prior use of medication to treat diabetes except gestational diabetes
* Use of drugs known to exacerbate glucose tolerance
* History of diabetes or prior use of medications to treat diabetes except GDM
* Creatinine clearance less than 60 ml/min
* Pregnancy planned during the coming two years
* Currently lactating
* Patient not willing to use adequate contraception during study period (unless sterilized)

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-09-28 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Elkind-Hirsch, Ph.D., Principal Investigator — Woman's Hospital, Louisiana; Martha Paterson, M.D., Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will only be shared with participant

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from November 2014 to September 2017. Patients were recruited from the Woman's Hospital Metabolic Clinic
Pre-assignment Details: . Patients were eligible for randomization if they had impaired fasting glucose (IFG), impaired glucose tolerance (IGT), or both (IFG/IGT) by OGTT. Patients with diabetes or normal glucose tolerance were excluded.
Groups:
- Sitagliptin-Metformin: 50 mg/1000 mg BID
  Sitagliptin-Metformin: Experimental -DPP-4 inhibitor- oral medication
Period: Overall Study
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Started | 12 | 12 | 12
Completed | 12 | 9 | 12
Not Completed | 0 | 3 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin | Total
Number analyzed (Participants) | 12 | 12 | 12 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 12 | 36
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Postpartum previous GDM females
  Participants
    Patients | 12 | 12 | 12 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 2 | 7
  White | 10 | 9 | 10 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 36
Hyperglycemia [Count of Participants; unit: Participants] | 12 | 12 | 12 | 36

OUTCOME MEASURES:

1. Primary Outcome: Normalization of Glucose Levels
Description: Normalization of glucose in patients with abnormal glucose levels is defined as a fasting glucose level of <100 mg/dL and a 2-hour glucose level following a 75 gram oral glucose load of <140 mg/dL
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Sitagliptin-Metformin: 50 mg/1000 mg twice a day (BID)
  Sitagliptin-Metformin: Experimental -DPP-4 inhibitor- oral medication
- Placebo Pill: 1 pill/ twice a day (BID) for 16 weeks
  Placebo pill: Will evaluate effect of lifestyle and diet only
- Metformin: 1000 mg twice a day (BID)
  Metformin: Biguanide- insulin sensitizer
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
Participants | 9 | 2 | 4
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Study change from dysglycemia to normal glucose state; Test type: Superiority; p = .035, McNemar

2. Secondary Outcome: Fasting Blood Glucose
Description: Blood glucose in the fasting state
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
mg/dL | 96 (13) | 101 (13) | 93 (6)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Subjects (SS)/ Treatment Group x repeated measures (visit) design; Test type: Superiority; p = 0.044, ANOVA

3. Secondary Outcome: Mean Blood Glucose Level From the Oral Glucose Tolerance Test (OGTT)
Description: The mean blood glucose is calculated by averaging the 4 blood glucose levels measure during a 75 gm oral glucose tolerance test . This involves summing the glucose levels measured at baseline, and 1/2 hour,1 hour and 2 hours after the glucose load and dividing by 4..
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
mg/dL | 113 (19) | 132 (17) | 143 (20)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.034, ANOVA

4. Secondary Outcome: Fasting Insulin Resistance
Description: Insulin resistance calculated from fasting glucose and insulin levels known as HOMA-IR
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
index | 2.4 (1.2) | 4.7 (3.8) | 2.6 (1.7)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = .047, ANOVA

5. Secondary Outcome: Matsuda Index of Insulin Sensitivity
Description: Composite insulin sensitivity index calculated from from glucose and insulin levels obtained during the OGTT
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
index | 6.2 (3.9) | 5.0 (4.9) | 5.2 (4)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.017, ANOVA

6. Secondary Outcome: Oral Disposition Index
Description: Measure of pancreatic beta cell compensatory action known as IS-SI
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
index | 427 (231) | 194 (93) | 170 (109)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.014, ANOVA

7. Secondary Outcome: Triglyceride/HDL-Cholesterol Ratio
Description: The ratio of triglyceride to HDL cholesterol is used as an indirect measure of insulin resistance
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
Ratio | 3.3 (1.4) | 4.5 (3.1) | 2.7 (1.5)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.042, ANOVA

8. Secondary Outcome: Body Mass Index
Description: Measure of body weight corrected by height
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: kg/meters^2
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
kg/meters^2 | 32.6 (8) | 33.5 (9) | 33.6 (6)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.002, ANOVA

9. Secondary Outcome: Waist Circumference
Description: Measure of central fat
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
centimeters | 90 (14) | 93 (17) | 93 (13)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.004, ANOVA

10. Secondary Outcome: Waist-to-Height Ratio
Description: Measure of central obesity adjusted for stature
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
Ratio | .54 (.09) | .57 (.1) | .58 (.07)
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Factorial repeated measures ANOVA with Bonferroni contrast test; Test type: Superiority; p = 0.004, ANOVA

11. Other Pre Specified Outcome: Liver Enzymes as Safety Measure
Description: Number of patients with no clinically significant changes in liver enzymes-measure of liver enzymes was a study safety endpoint
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
Number analyzed (Participants) | 12 | 9 | 12
Participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Sitagliptin-Metformin vs Placebo Pill vs Metformin; Test type: Superiority; p = 0.9, Fisher Exact

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Sitagliptin-Metformin | Placebo Pill | Metformin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 0/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin-Metformin (N=12) | Placebo Pill (N=12) | Metformin (N=12)
Diarrhea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 3 (4)

LIMITATIONS AND CAVEATS:
Important limitations of the present study were the small number of patients in the treatment groups and the short interval (16 weeks) of drug treatment. Second, surrogate measures were used to estimate insulin sensitivity and secretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT01856907/Prot_SAP_000.pdf